CLINICAL TRIAL: NCT04923360
Title: Morphological Parameters of Blood Cell's Activation in Characterization and Prognosis in a COPD Patients Cohort
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Galdakao-Usansolo (Other Government)
Collaborators: Osakidetza (Other)
Responsible Party: Principal Investigator, Dr. Cristobal Esteban, MD, Hospital Galdakao-Usansolo
Other Study IDs: G95756334
Record Dates: First submitted 2021-04-11; First posted 2021-06-11 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-04

CONDITIONS: COPD
Keywords: COPD prognostic; COPD characterization; Cellular Popular Data
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Inflammation markers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Though exacerbations in the COPD (Chronic Pulmonary Obstructive Disease) and specially the most severe cases (hospitalizations) are currently a fundamental outcome in the COPD due to its clinical and economic significance, there are many unanswered questions still today such as the very definition of exacerbation itself.

Research parameters like the CPD (Cell Population Data) are added to the basic blood count. The CPD of the XN analyzers (Sysmex Corporation, Kobe, Japan) provide quantitative information of the morphological and functional characteristics of the leukocytes: their volume, content of nucleic acids and structure of the cytoplasm. The CPD are numerical data which represent the morphology which characterizes the neutrophils, lymphocytes, monocytes, eosinophils and platelets classifying them as per their volume and shape, granularity and their content of nucleic acids. The approach is that such cheap and accessible technique can provide relevant information in the area of COPD exacerbations.

Therefore, this study proposes several objectives:

1. Establish the CPD values for each phenotype of COPD (both for those already established in the Spanish guide of COPD and in the potential phenotypes which may be established in this study based on the CPDs themselves).
2. Identify which, among the CPDs, are more relevant in relation to cellular activation (neutrophils, lymphocytes, eosinophils and platelets) both in the stage of clinical stability and during the severe exacerbation.
3. Establish different phenotypes of COPD (in stable phase) according to the CPD values.
4. Determine the existence of an association between the level of activation of these cells in stability phase of the COPD and the risk of exacerbation; establish the optimum cutoff points.

The study will include 500 patients with different levels of COPD in the OSI-Barrualde and OSI-Bilbao. Several clinical measurements will be carried out for their characterization. CPD measurements will be made both in clinical stability phase or during exacerbations.

DETAILED DESCRIPTION:
One of the most analyzed outcomes in COPD (Chronic Pulmonary Obstructive Disease) are the exacerbations, specially the severe ones. There are two challenges in relation to severe exacerbations: one related to the high use of sanitary resources and costs; and the second one, related to the worsening of the pulmonary function and the quality of life.

Nowadays in the Spanish COPD guideline called GESEPOC (Guía Española de la Enfermedad Pulmonar Obstructiva Crónica), there is a COPD "exacerbator" phenotype. However, there are some limitations round the COPD exacerbation, like its definition or its predictors. In other words, there are no indicators that can help the investigators to define more precisely an exacerbation or the COPD exacerbator profile.

COPD is a chronic disease with low intensity, systemic and chronic inflammation. The matter is that it is not established which indicators the investigators have to use to determinate it. There are some indicators like C reactive protein, TNF-alpha, IL-6 (Interleukin 6), microalbumins and adiponectin; and there are also prognostic scores based on them. However, they cannot help the investigators to establish COPD phenotypes of patients that can suffer an exacerbation. The investigators neither have indicators in stable phase that say them the risk of an exacerbation. Moreover, it is said that there are different types of exacerbations and even it has been established indicators of these exacerbation phenotypes. However, nowadays it cannot be translated into daily clinical practice. If investigators would be able to do it, they could advance in the knowledge of the exacerbations and they could establish precision treatments.

The blood count is one of the most required laboratory test in clinical practice. It is cost-effective because of its low price and the huge quantity of information it brings. After adapting the flow cytometry in hematologic modern analyzers, a more detailed study of cells can be done. Moreover, morphological changes can be detected in response to different stimulus, like infections or the ones that are caused by inflammatory reactions.

In this project, CPD ("Cellular Popular Data") is added to the basis blood count. They are parameters that are under investigation nowadays. The CPD of the XN analyzers (Sysmex Corporation, Kobe, Japan) give quantitative information about morphological and functional characteristics of leukocytes: their volume, the quantity of nucleic acid they contain and the structure of the cytoplasm. The CPD are numeric data that represent the morphology of the neutrophils, lymphocytes, monocytes and eosinophils, and they classify them by their volume, form, granularity and nucleic acid content. The same technology allows to the analyzer to classify the platelets by their morphology, what is related to its thrombogenic activity.

The composition of the membrane of the activated cells is different from the one of cells that are at rest, because of the expression of the receptors and the surface signaling molecules, in response to the activation. This membrane is more sensitive to the reagents of the analyzer, and more quantity of fluorescent colorant can enter in the activated cell and link to the cytoplasmic organelles and nucleic acids. The optic signals are different, what allows to distinguish morphological changes, and they are directly related to the cell functionality.

The activated neutrophils and monocytes have more "deformability", mobility and more capacity to adhesion, granulation and liberation of cytokines.

CPD values reflect morphological and functional transformation of these activated cells, and they give us very important information of the state of the cell and the state of the patient at the moment the sample is taken.

In addition, CPD support the differentiation between viral and bacterial infections or between acute and chronic infections, but also they say if there is an inflammatory condition without infection, with better diagnostic performance than conventional parameters, like total leukocytes, neutrophiles percentage and C reactive protein, that traditionally are used like acute infection markers.

Currently available literature speaks about the utility of CPD in the diagnosis, but there is no data about their possible prognostic value.

Respect from blood cells, previous COPD studies showed the relation between neutrophils/lymphocytes and platelets/lymphocytes as prognostic factors during severe exacerbations in COPD. Nowadays, it is emphasized the importance of eosinophils in COPD like predictor of exacerbation, like exacerbation severity marker and like response marker to the treatment in stable and in the exacerbation phase. It is thought that in this study the prognostic capacity of these new approaches can be better, becauseit is included the grade of activation of these cells like key parameter. This is a novel approach in the COPD field.

On the other hand, other inflammatory biomarkers (TNF-alpha, IL-6…) are expensive and less accessible in the daily clinical practice, while the evaluation of these new biomarkers of leukocytes are cheaper and more available in routine clinical practice by the blood count.

These new biomarkers could help the investigators confirming the inflammatory response and recognizing patients that could exacerbate. They also could determine the kind of their exacerbation and their prognosis.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis following American Thoracic Association (Am Rev Respir Dis 1987;136:225-244), FEV1/FVC < 70% (FEV1: forced expiratory volume in one second, FVC: forced vital capacity) post-bronchodilator. Acceptation to participate in the study by the informed consent.

Exclusion Criteria:

* Concomitant diseases that could interfere in the realization of the measures in the study (dementia, severe psychiatric disease, invalidating neurological diseases, important deafness, active neoplasms); patients with asthma as main diagnostic; patients with bronchiectasis as main disease or with extensive sequels of pulmonary tuberculosis; patients that in the beginning seem to be unable to follow the procedures of the study (questionnaires, pulmonary function test, 6 minutes walking test…); patients with difficulties to walk; patients with active infections or chronic inflammatory diseases; patients that reuse to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COPD diagnosis following American Thoracic Association (Am Rev Respir Dis 1987;136:225-244), FEV1/FVC < 70% post-bronchodilator. The diagnosis of COPD and the treatment must be at least 6 months before the inclusion in the study.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Establish CPD (Cellular Popular Data) values for each phenotype of COPD. | 3 years
  * CPD (Cellular Popular Data): morphological parameters measured in the blood count cells (neutrophils, lymphocytes, eosinophils and platelets).
  * Phenotypes of COPD described in Spanish COPD guideline (GesEPOC):
  * No exacerbator: patient with 0-1 exacerbation per year, without admission
  * Exacerbator with emphysema: patient with emphysema and 2 or more exacerbations per year or 1 admission
  * Exacerbator with chronic bronchitis: patient with chronic bronchitis and 2 or more exacerbations per year or 1 admission
  * Mixed phenotype: asthma-COPD overlap: a patient with COPD and diagnostic criteria for asthma, or with a very positive bronchodilator test (increase in FEV1> 400ml and 15%) and / or peripheral blood eosinophilia greater than 300cells / mm3.

SECONDARY OUTCOMES:
Identify which, among the CPDs, are more relevant in relation to cellular activation (neutrophils, lymphocytes, eosinophils and platelets) both in the stage of clinical stability and during the severe exacerbation. | 3 years
  * CPD (Cellular Popular Data): morphological parameters measured in the blood count cells (neutrophils, lymphocytes, eosinophils and platelets).
  * To define clinical status:
  * Evaluation of dyspnea: mMRC (Modified Medical Research Council) scale Dyspnea only with strenuous exercise: 0 Dyspnea when hurrying or walking up a slight hill: 1 Walks slower than people of the same age because of dyspnea or has to stop for breath when walking at own pace: 2 Stops for breath after walking 100 yards (91 m) or after a few minutes: 3 Too dyspneic to leave house or breathless when dressing: 4
  * Functional respiratory examination (flow-volume curve, lung volumes, diffusing capacity of the lungs for carbon monoxide (DLCO).
  * Exercise capacity (6 minute walking test)
  * Inflammation markers (C reactive protein, TNF-alpha, IL-6 (Interleukin 6), IL-1 (Interleukin 1), IL-8 (Interleukin 8), IGF-I and adiponectin).
  * Sputum culture.
Establish new phenotypes of COPD | 3 years
  * CPD (Cellular Popular Data): morphological parameters measured in the blood count cells (neutrophils, lymphocytes, eosinophils and platelets).
  * Clinical status is described in previous outcome.
Determine the existence of an association between the level of activation of these cells in stability phase of COPD and the risk of exacerbation | 3 years
  * CPD (Cellular Popular Data): morphological parameters measured in the blood count cells (neutrophils, lymphocytes, eosinophils and platelets).
  * Clinical status is described in previous outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Cristobal Esteban, MD, Principal Investigator — Osakidetza
Locations (1):
- Hospital Galdakao Usansolo, Galdakao, Vizcaya, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mathers CD, Loncar D. Projections of global mortality and burden of disease from 2002 to 2030. PLoS Med. 2006 Nov;3(11):e442. doi: 10.1371/journal.pmed.0030442. PMID 17132052
- [Background] World Health Organization. Chronic Obstructive Pulmonary Disease (COPD). Avalaible from: http:// www.who.int/respiratory/copd/en/index.html
- [Background] Donaldson GC, Seemungal TA, Bhowmik A, Wedzicha JA. Relationship between exacerbation frequency and lung function decline in chronic obstructive pulmonary disease. Thorax. 2002 Oct;57(10):847-52. doi: 10.1136/thorax.57.10.847. PMID 12324669
- [Background] Esteban C, Quintana JM, Moraza J, Aburto M, Egurrola M, Espana PP, Perez-Izquierdo J, Aguirre U, Aizpiri S, Capelastegui A. Impact of hospitalisations for exacerbations of COPD on health-related quality of life. Respir Med. 2009 Aug;103(8):1201-8. doi: 10.1016/j.rmed.2009.02.002. Epub 2009 Mar 9. PMID 19272762
- [Background] Soler-Cataluna JJ, Martinez-Garcia MA, Roman Sanchez P, Salcedo E, Navarro M, Ochando R. Severe acute exacerbations and mortality in patients with chronic obstructive pulmonary disease. Thorax. 2005 Nov;60(11):925-31. doi: 10.1136/thx.2005.040527. Epub 2005 Jul 29. PMID 16055622
- [Background] Yoon HI, Li Y, Man SFP, Tashkin D, Wise RA, Connett JE, Anthonisen NA, Churg A, Wright JL, Sin DD. The complex relationship of serum adiponectin to COPD outcomes COPD and adiponectin. Chest. 2012 Oct;142(4):893-899. doi: 10.1378/chest.11-2173. PMID 22207678
- [Background] Romundstad S, Naustdal T, Romundstad PR, Sorger H, Langhammer A. COPD and microalbuminuria: a 12-year follow-up study. Eur Respir J. 2014 Apr;43(4):1042-50. doi: 10.1183/09031936.00160213. Epub 2014 Jan 16. PMID 24435009
- [Background] Zemans RL, Jacobson S, Keene J, Kechris K, Miller BE, Tal-Singer R, Bowler RP. Multiple biomarkers predict disease severity, progression and mortality in COPD. Respir Res. 2017 Jun 13;18(1):117. doi: 10.1186/s12931-017-0597-7. PMID 28610627
- [Background] Garcia-Rivero JL, Esquinas C, Barrecheguren M, Bonnin-Vilaplana M, Garcia-Sidro P, Herrejon A, Martinez-Rivera C, Malo de Molina R, Marcos PJ, Mayoralas S, Naval E, Ros JA, Valle M, Miravitlles M. Risk Factors of Poor Outcomes after Admission for a COPD Exacerbation: Multivariate Logistic Predictive Models. COPD. 2017 Apr;14(2):164-169. doi: 10.1080/15412555.2016.1260538. Epub 2016 Dec 16. PMID 27983876
- [Background] Bafadhel M, McKenna S, Terry S, Mistry V, Reid C, Haldar P, McCormick M, Haldar K, Kebadze T, Duvoix A, Lindblad K, Patel H, Rugman P, Dodson P, Jenkins M, Saunders M, Newbold P, Green RH, Venge P, Lomas DA, Barer MR, Johnston SL, Pavord ID, Brightling CE. Acute exacerbations of chronic obstructive pulmonary disease: identification of biologic clusters and their biomarkers. Am J Respir Crit Care Med. 2011 Sep 15;184(6):662-71. doi: 10.1164/rccm.201104-0597OC. PMID 21680942
- [Background] Arostegui I, Esteban C, Garcia-Gutierrez S, Bare M, Fernandez-de-Larrea N, Briones E, Quintana JM; IRYSS-COPD Group. Subtypes of patients experiencing exacerbations of COPD and associations with outcomes. PLoS One. 2014 Jun 3;9(6):e98580. doi: 10.1371/journal.pone.0098580. eCollection 2014. PMID 24892936
- [Background] Linssen J, Aderhold S, Nierhaus A, Frings D, Kaltschmidt C, Zanker K. Automation and validation of a rapid method to assess neutrophil and monocyte activation by routine fluorescence flow cytometry in vitro. Cytometry B Clin Cytom. 2008 Sep;74(5):295-309. doi: 10.1002/cyto.b.20422. PMID 18431775
- [Background] Cornet E, Boubaya M, Troussard X. Contribution of the new XN-1000 parameters NEUT-RI and NEUT-WY for managing patients with immature granulocytes. Int J Lab Hematol. 2015 Oct;37(5):e123-6. doi: 10.1111/ijlh.12372. Epub 2015 Apr 28. No abstract available. PMID 25923650
- [Background] Buoro S, Seghezzi M, Vavassori M, Dominoni P, Apassiti Esposito S, Manenti B, Mecca T, Marchesi G, Castellucci E, Azzara G, Ottomano C, Lippi G. Clinical significance of cell population data (CPD) on Sysmex XN-9000 in septic patients with our without liver impairment. Ann Transl Med. 2016 Nov;4(21):418. doi: 10.21037/atm.2016.10.73. PMID 27942509
- [Background] Urrechaga E, Boveda O, Aguirre U. Role of leucocytes cell population data in the early detection of sepsis. J Clin Pathol. 2018 Mar;71(3):259-266. doi: 10.1136/jclinpath-2017-204524. Epub 2017 Aug 18. PMID 28821583
- [Background] Kaeslin M, Brunner S, Raths J, Huber A. Improvement in detecting bacterial infection in lower respiratory tract infections using the Intensive Care Infection Score (ICIS). J Lab Med 2016; 40: 175-182.
- [Background] Zhu Y, Cao X, Tao G, Xie W, Hu Z, Xu D. The lymph index: a potential hematological parameter for viral infection. Int J Infect Dis. 2013 Jul;17(7):e490-3. doi: 10.1016/j.ijid.2012.12.002. Epub 2013 Jan 10. PMID 23313156
- [Background] Henriot I, Launay E, Boubaya M, Cremet L, Illiaquer M, Caillon H, Desjonqueres A, Gillet B, Bene MC, Eveillard M. New parameters on the hematology analyzer XN-10 (SysmexTM) allow to distinguish childhood bacterial and viral infections. Int J Lab Hematol. 2017 Feb;39(1):14-20. doi: 10.1111/ijlh.12562. Epub 2016 Aug 30. PMID 27572612
- [Background] Xu D. Clinical Applications of Leukocyte Morphological Parameters Int J Pathol Clin Res 2015; 1:002
- [Background] Yao C, Liu X, Tang Z. Prognostic role of neutrophil-lymphocyte ratio and platelet-lymphocyte ratio for hospital mortality in patients with AECOPD. Int J Chron Obstruct Pulmon Dis. 2017 Aug 3;12:2285-2290. doi: 10.2147/COPD.S141760. eCollection 2017. PMID 28814856
- [Background] Paliogiannis P, Fois AG, Sotgia S, Mangoni AA, Zinellu E, Pirina P, Negri S, Carru C, Zinellu A. Neutrophil to lymphocyte ratio and clinical outcomes in COPD: recent evidence and future perspectives. Eur Respir Rev. 2018 Feb 7;27(147):170113. doi: 10.1183/16000617.0113-2017. Print 2018 Mar 31. PMID 29436405
- [Background] Bafadhel M, Pavord ID, Russell REK. Eosinophils in COPD: just another biomarker? Lancet Respir Med. 2017 Sep;5(9):747-759. doi: 10.1016/S2213-2600(17)30217-5. Epub 2017 Jun 7. PMID 28601554
- [Background] Kerkhof M, Sonnappa S, Postma DS, Brusselle G, Agusti A, Anzueto A, Jones R, Papi A, Pavord I, Pizzichini E, Popov T, Roche N, Ryan D, Thomas M, Vogelmeier C, Chisholm A, Freeman D, Bafadhel M, Hillyer EV, Price DB. Blood eosinophil count and exacerbation risk in patients with COPD. Eur Respir J. 2017 Jul 20;50(1):1700761. doi: 10.1183/13993003.00761-2017. Print 2017 Jul. No abstract available. PMID 28729477
- [Background] Vedel-Krogh S, Nielsen SF, Lange P, Vestbo J, Nordestgaard BG. Blood Eosinophils and Exacerbations in Chronic Obstructive Pulmonary Disease. The Copenhagen General Population Study. Am J Respir Crit Care Med. 2016 May 1;193(9):965-74. doi: 10.1164/rccm.201509-1869OC. PMID 26641631
- [Background] Pascoe S, Locantore N, Dransfield MT, Barnes NC, Pavord ID. Blood eosinophil counts, exacerbations, and response to the addition of inhaled fluticasone furoate to vilanterol in patients with chronic obstructive pulmonary disease: a secondary analysis of data from two parallel randomised controlled trials. Lancet Respir Med. 2015 Jun;3(6):435-42. doi: 10.1016/S2213-2600(15)00106-X. Epub 2015 Apr 12. PMID 25878028